CLINICAL TRIAL: NCT03892902
Title: A Single-center, Randomized, Double-blind, Double-dummy, Placebo- and Active-controlled, 4-way Cross-over Study to Assess Next-day Driving Performance Following Single and Multiple Evening Administrations of ACT-541468 in Middle-aged and Elderly Subjects
Brief Title: A Clinical Study to Assess Next-day Driving Performance Following Administration of ACT-541468 in Middle-aged and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-078-108
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant; zopiclone

STUDY DESIGN:
Intervention Model Description: 4-way cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (50 mg ACT-541468) (Experimental): 1 tablet of ACT-541468 50 mg + 1 tablet of ACT-541468 matching placebo + zopiclone matching placebo administered in the evening on Days 1-4 of Treatment Period A.
  Interventions: Drug: ACT-541468; Other: Placebo
- Treatment B (100 mg ACT-541468) (Experimental): 2 tablets of ACT-541468 50 mg + zopiclone matching placebo administered in the evening on Days 1-4 of Treatment Period B.
  Interventions: Drug: ACT-541468; Other: Placebo
- Treatment C (7.5 mg zopiclone) (Experimental): 2 tablets of ACT-541468 matching placebo + 1 capsule of zopiclone 7.5 mg administered in the evening on Days 1 and 4 of Treatment Period C. In the evenings of Days 2 and 3, subjects will receive placebo (i.e., 2 tablets of ACT-541468 matching placebo + zopiclone matching placebo).
  Interventions: Drug: Zopiclone 7.5 mg; Other: Placebo
- Treatment D (placebo) (Experimental): 2 tablets of ACT-541468 matching placebo + zopiclone matching placebo administered in the evening on Days 1-4 of Treatment Period D.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ACT-541468 — Film-coated tablet for oral use at a dose strength of 50 mg.
  Arms: Treatment A (50 mg ACT-541468); Treatment B (100 mg ACT-541468)
Drug: Zopiclone 7.5 mg — Over-encapsulated to maintain blinding.
  Arms: Treatment C (7.5 mg zopiclone)
Other: Placebo — Matching to maintain blinding.

SUMMARY:
A clinical study to assess next-day driving performance following evening administrations of ACT-541468 in middle-aged and elderly subjects

ELIGIBILITY:
Inclusion Criteria

General criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male and female subjects aged between 50 and 80 years (inclusive) at Screening.
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 pre-dose of each treatment period. They must consistently and correctly use a highly effective method of contraception, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential (i.e., postmenopausal, XY genotype, Turner syndrome, uterine agenesis).

Study-specific criteria

* Subject has a valid driving license for more than 5 years, has driven at least 3000 km/year on average in the past 2 years.
* Normal visual acuity (corrected or uncorrected).

Exclusion Criteria:

General criteria:

* Pregnant or lactating women.
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results.
* History or presence of rhythm disorders
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Study-specific criteria:

* Current or previous diagnosis of insomnia-related disorder according to the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria.
* History of alcoholism, drug abuse, or regular use of sedative drugs or hypnotics within 3 years prior to Screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of more than 21 units or an average daily intake of more than 3 units (males), or defined as an average weekly intake of more than 14 units or an average daily intake of more than 2 units (females). One unit is equivalent to a half-pint (approx. 250 mL) of beer or 1 measure (25 mL) of spirits or 1 glass (125 mL) of wine.
* Modified Swiss Narcolepsy Scale total score < 0 at Screening or history of narcolepsy or cataplexy.
* Activities that disturb the circadian rhythm (e.g., working night shift, travelling across 3 time zones) within 2 weeks before (each) study treatment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic endpoint: Driving performance as measured by the SDLB (difference from placebo, cm) using the Green Dino driving simulator - Day 2 | On Day 2 at 9 hours post dose. Duration of the test: 1 hour
  SDLP = standard deviation of the lateral position
Pharmacodynamic endpoint: Driving performance as measured by the SDLB (difference from placebo, cm) using the Green Dino driving simulator - Day 5 | On Day 5 at 9 hours post dose. Duration of the test: 1 hour
  SDLP = standard deviation of the lateral position

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Pharmacologist, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No